CLINICAL TRIAL: NCT04332588
Title: Monitoring HER2+ Breast Cancer Neoadjuvant Treatment With Advanced PET/MRI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, Director, Advanced Imaging Facility, Director, Division of Molecular Imaging and Therapeutics Professor, Division of Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 300005387; O'Neal Invests Award (Other: UAB O'Neal Comprehensive Cancer Center)
Record Dates: First submitted 2020-03-23; First posted 2020-04-02 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Herceptin monotherapy cohort (Experimental): Herceptin monotherapy cohort. Locally advanced HER2+ breast cancer patients receiving neoadjuvant Herceptin monotherapy prior to combination therapy will undergo three contrast-enhanced [18F]FMISO PET/MRI scans. Each imaging session will be identical. Imaging session one will be after diagnosis and before beginning monotherapy. Imaging session two will be within 10 days prior to beginning combination therapy with targeted HER2 agents. Imaging session three will be within 10 days prior to beginning the second round of combination therapy with targeted HER2 agents.
  Interventions: Drug: [18F]FMISO PET/MRI imaging
- Combination therapy cohort (Experimental): Locally advanced HER2+ breast cancer patients that receiving neoadjuvant combination therapy including Herceptin will undergo two contrast-enhanced [18F]FMISO PET/MRI imaging. Imaging session one will be after diagnosis and before beginning combination therapy. Imaging session two will be within 10 days prior to beginning the second round of combination therapy with targeted HER2 agents.
  Interventions: Drug: [18F]FMISO PET/MRI imaging

INTERVENTIONS:
Drug: [18F]FMISO PET/MRI imaging — [18F]FMISO PET/MRI imaging

SUMMARY:
The purpose of the study is to see if using an investigational drug called [18F]FMISO with PET/MRI imaging can help monitor and predict the effect of trastuzumab (Herceptin) on chemotherapy in patients diagnosed with advanced HER2 positive breast cancer. This study is for imaging purposes only and is not a treatment study. The results of this study will not change a patient's clinical treatment plan but it may help physicians and researchers better understand how best to treat patients with breast cancer in the future.

DETAILED DESCRIPTION:
There are 2 groups or cohorts in this study. The cohort patient's are in is based on their clinical treatment plan set by your physician. The number of imaging visits and timing of visits will be determined by what cohort they are in.

If the patient is in cohort #1, they will make 4 visits to UAB. They will be scheduled for a pre-study or screening visit. During the pre-study visit, once consented, they will have a blood draw to determine kidney function, and a pregnancy test if they are a woman of childbearing potential. Their vital signs will be taken, they will be asked to fill out an MRI questionnaire, and they will have a PET/MRI fit test. If eligible for the study, they will be scheduled for the first PET imaging visit which will occur before they start chemotherapy. During this PET imaging visit, they will have a pregnancy test if they are a woman of childbearing potential. A plastic catheter will be placed into a vein in their arm and they will then be positioned in the PET/MRI scanner. Once positioned, they will be injected with the investigational radioactive drug, [18F]FMISO. They will then be imaged for up to 90 minutes during which time they will receive an FDA approved contrast agent called Prohance (gadoteridol). Once all the procedures are complete, the catheter will be removed and they may resume all normal activities. The patient will receive a follow-up phone call within 24-48 hours of your injection to be sure they are not experiencing any adverse events. Their second imaging visit will be scheduled after they receive therapy with Herceptin alone and within 10 days before their first cycle of combination therapy including Herceptin. During the second PET imaging visit, the same procedures will be followed as were performed during your first PET imaging visit. They will receive a follow-up phone call within 24-48 hours of your injection to be sure you are not experiencing any adverse events. Their third PET imaging visit will be scheduled after their first cycle of combination therapy including Herceptin and within 10 days before starting their second cycle of combination therapy including Herceptin. During the third PET imaging visit, the same procedures will be followed as were performed during their first and second PET imaging visits. The patient will receive a follow-up phone call within 24-48 hours of their injection to be sure they are not experiencing any adverse events.

If the patients are in cohort #2, they will make 3 visits to UAB. The patients will be scheduled for a pre-study or screening visit. During the pre-study visit, once consented, they will have a blood draw to determine kidney function, and a pregnancy test if they are a woman of childbearing potential. Their vital signs will be taken, they will be asked to fill out an MRI questionnaire, and they will have a PET/MRI fit test. If eligible for the study, they will be scheduled for the first PET imaging visit which will occur before they start chemotherapy. During this visit, they will have a pregnancy test if they are a woman of childbearing potential. A plastic catheter will be placed into a vein in their arm and they will then be positioned in the PET/MRI scanner. Once positioned, the patient will be injected with the investigational radioactive drug, [18F]FMISO. They will then be imaged for up to 90 minutes during which time they will receive an FDA approved contrast agent called Prohance (gadoteridol). Once all the procedures are complete, the catheter will be removed and the patient may resume all normal activities. They will receive a follow-up phone call within 24-48 hours of your injection to be sure they are not experiencing any adverse events. Your second PET imaging visit will be scheduled after your first cycle of combination therapy including Herceptin and within 10 days before starting the second cycle of combination therapy including Herceptin. During the third PET imaging visit, the same procedures will be followed as were performed during the first PET imaging visits. The patient will receive a follow-up phone call within 24-48 hours of your injection to be sure they are not experiencing any adverse events.

We will follow the patients every 6 months for 5 years by reviewing their medical records to see how they are doing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 18 years old and ≤ 75 years old
2. HER2+ breast cancer determined on primary tumor by a local pathology laboratory and defined as IHC score 3+ and/or positive by ISH (defined by ISH ratio of ≥ 2.0 for the number of HER2 gene copies to the number of chromosome 17 copies). Only one positive result is required for eligibility
3. Locally advanced stage II-III HER2+ breast cancer patients eligible for neoadjuvant therapy who are naïve to beginning treatment
4. Estimated life expectancy of greater than one year
5. Patients must have one lesion with RECIST measurable disease (great than 1 cm in diameter)

Exclusion Criteria:

1. Inability to provide informed consent F
2. Weight over 350 lbs., due to the scanner bore size
3. Lactating, known or suspected pregnancy. Women with child-bearing potential must a have a negative serum β-hCG pregnancy test within 48 hours or a negative urine β-hCG pregnancy test within 48 hours of each PET imaging study.
4. Contraindication for MRI study (e.g. non-removable metal implants or certain tattoos)
5. Unable to lie still on the imaging table for one (1) hour
6. contraindication for gadolinium-based contrast agent, ProHance (gadoteridol)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Baseline measure of PET standardized uptake value (SUV). | Baseline
  Compare baseline metrics from PET/MRI
Baseline measure of apparent diffusion coefficient (ADC) in mm2/sec from MRI. | Baseline
  Compare baseline metrics from PET/MRI
Baseline measure of signal enhancement ratio (SER) from MRI. | Baseline
  Compare baseline metrics from PET/MRI
Changes in SER from MRI | Baseline through 6 months
  Compare percent change of SER from imaging visit 3 to the baseline.
Changes in ADC from MRI | Baseline through 6 months
  Compare percent change of ADC (mm2/sec) from imaging visit 3 to the baseline.
Changes in SUV from PET | Baseline through 6 months
  Compare percent change of SUV from imaging visit 3 to the baseline.

SECONDARY OUTCOMES:
Follow-up | Baseline through 5 years
  Compare changes in imaging metrics to neoadjuvant response (defined as pathological complete response, near-pathological response, residual disease).
Follow-up | Baseline through 5 years
  Compare changes in imaging metrics to clinical response (defined as disease free-survival or recurrence).
Changes in ADC (mm2/sec) from MRI. | Baseline through 2 months
  Compare percent change from imaging visit 2 to the baseline.
Changes in SER from MRI. | Baseline through 2 months
  Compare percent change from imaging visit 2 to the baseline.
Changes in SUV from PET. | Baseline through 2 months
  Compare percent change from imaging visit 2 to the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan McConathy, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States